CLINICAL TRIAL: NCT02527005
Title: A Comparative Study of Azithromycin and Sulphadoxine-pyrimethamine as Prophylaxis Against Malaria in Pregnant HIV Positive Patients
Brief Title: A Comparative Study of Azithromycin and S-P as Prophylaxis in Pregnant HIV+ Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, ORIYOMI OMOTOYOSI AKINYOTU, Senior Registrar, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UIbadan
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Malaria; Pregnant; HIV
Keywords: IPT; malaria; pregnant; HIV positive
MeSH Terms: conditions — Malaria; HIV Seropositivity | interventions — fanasil, pyrimethamine drug combination; Azithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Active Comparator): Tabs Azithromycin 500mg daily for 3 days
  Interventions: Drug: Sulphadoxine-pyrimethamine; Drug: Azithromycin
- Sulphadoxine-pyrimethamine (Active Comparator): 500mg of sulphadoxine and 25mg of pyrimethamine 3 tablets every 4 weeks for 3 doses
  Interventions: Drug: Sulphadoxine-pyrimethamine; Drug: Azithromycin

INTERVENTIONS:
Drug: Sulphadoxine-pyrimethamine — Sulphadoxine-Pyrimethamine 500mg of Sulphadoxine and 25mg of Pyrimethamine 3tablets monthly for 3 doses
  Other Names: Vitadar
Drug: Azithromycin — Tabs Azithromycin 500mg daily for 3 days
  Other Names: Zithromax

SUMMARY:
Randomized controlled single blind prospective comparative study

DETAILED DESCRIPTION:
This study is intended to be a randomized controlled single blind prospective comparative study conducted to compare the efficacy of three monthly doses of sulphadoxine-pyrimethamine as intermittent preventive therapy for malaria with azithromycin in HIV positive pregnant women

ELIGIBILITY:
Inclusion Criteria:

* Pregnant HIV positive patients,
* Gestational age 16 weeks and above,
* No history of azithromycin or sulphadoxine-pyrimethamine use four weeks prior to recruitment

Exclusion Criteria:

* Anaemia packed cell volume less than 30%,
* pre-existing medical conditions- diabetes mellitus,
* hypertension,
* allergy to sulphadoxine-pyrimethamine or azithromycin

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Level of malaria parasitemia at delivery in HIV positive women following administration of Azithromycin or Sulphadoxine- pyrimethamine as intermittent preventive therapy for malaria in pregnancy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: AYODELE O AROWOJOLU, MBBS IBADAN, Study Director — UNIVERSITY COLLEGE HOSPITAL,IBADAN,OYO STATE, NIGERIA; ORIYOMI O AKINYOTU, MBBS IBADAN, Principal Investigator — UNIVERSITY COLLEGE HOSPITAL, IBADAN, OYO STATE, NIGERIA; ADENIKE F BELLO, MBBS IBADAN, Study Director — UNIVERSITY COLLEGE HOSPITAL, IBADAN, OYO STATE, NIGERIA; ADEOLA R ABDUS-SALAM, MBBS IBADAN, Study Director — ADEOYO MATERNITY TEACHING HOSPITAL, IBADAN, OYO STATE
Locations (1):
- University College Hospital,, Ibadan, Oyo State, Nigeria

REFERENCES:
- [Background] Taylor WR, Richie TL, Fryauff DJ, Picarima H, Ohrt C, Tang D, Braitman D, Murphy GS, Widjaja H, Tjitra E, Ganjar A, Jones TR, Basri H, Berman J. Malaria prophylaxis using azithromycin: a double-blind, placebo-controlled trial in Irian Jaya, Indonesia. Clin Infect Dis. 1999 Jan;28(1):74-81. doi: 10.1086/515071. PMID 10028075
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693